CLINICAL TRIAL: NCT06032273
Title: Exploring Caregiver Needs While Supporting People with CF Learning About Lung Transplant
Brief Title: Lung Transplant READY CF 2: CARING CF Ancillary RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Principal Investigator, Kathleen Ramos, Associate Professor, Division of Pulmonary, Critical Care and Sleep Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: STUDY00016943
Record Dates: First submitted 2023-08-26; First posted 2023-09-11 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Lung Transplantation; Advanced Lung Disease; Caregiver
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Access to investigator-designed lung transplant education website (Experimental): Access to an investigator-designed web-based educational resource with information about lung transplant for three months.
  Interventions: Behavioral: Investigator-designed lung transplant education website
- No access to lung transplant education website (No Intervention): No access to the investigator-designed lung transplant educational resource.

INTERVENTIONS:
Behavioral: Investigator-designed lung transplant education website — Caregiver participants assigned to the intervention will access the investigator-designed educational resource via their login to a secure website.
  Arms: Access to investigator-designed lung transplant education website

SUMMARY:
Lung transplant is an option for treating end-stage lung disease in cystic fibrosis (CF). In the United States, more people with CF and low lung function die each year than undergo lung transplant. More than half of people with CF who die without a lung transplant were never referred for consideration. Patient preference not to undergo lung transplant may account for 25-40% of decisions to defer referral.

Patients' health discussion networks function to support individuals in health related matters and may provide critical support during the lung transplant journey. Increasing awareness of lung transplant, and promoting the process of deliberation and utilization of social support, could reduce the number of people with CF who die without lung transplant. Additionally, the most common patient-endorsed barrier to lung transplant discussions is a worry about being a burden on family and friends after lung transplant. For lung transplant recipients with complex post-operative courses, low social support is associated with increased mortality. Additionally, adequate social support is a requirement at all lung transplant programs in the US.

Investigators are interested in understanding how caregivers may benefit from using lung transplant educational resources and how caregivers prepare for having discussions with their loved ones and/or helping them make decisions about lung transplant as a treatment option for advanced CF. The purpose of this study is to test whether an investigator-designed research website compared to no caregiver intervention reduces caregiver burden (assessed with the Brief Assessment Scale for Caregivers, BASC), caregiver preparedness for lung transplant discussions, and caregiver lung transplant knowledge as an ancillary study in a multicenter RCT. Further, investigators will assess patient perceptions of caregiver support as measured by the Social Support Effectiveness Questionnaire (SSE-Q) and evaluate caregivers' willingness to provide support through semi-structured interviews in patient-caregiver dyads.

Study involvement will span 6 months and study activities will involve the following:

* Three Zoom research sessions (15-90 minutes each)
* Survey assessments and an interview
* Access to a research website that contains educational resources about lung transplant

DETAILED DESCRIPTION:
Lung transplant is an option for treating end-stage lung disease in cystic fibrosis (CF). In the US, more CF patients with forced expiratory volume in 1 second (FEV1) less than 30% of predicted die each year than undergo lung transplant. More than half of patients who die without lung transplant were never referred for consideration. This is especially relevant for disproportionately impacted communities with limited access to lung transplant ("communities of concern"), including patients of lower socioeconomic status, minoritized race (e.g. Black, Asian), or Hispanic ethnicity. Patient preference may account for 25-40% of decisions to defer referral, but may at times be informed by inaccurate assumptions. Patients' health discussion networks function to support individuals in health related matters and may provide critical support during the lung transplant journey. Increasing awareness of lung transplant, and promoting the process of deliberation and utilization of social support, could reduce the number of people with CF who die without lung transplant. The CF Foundation (CFF) lung transplant referral guidelines recommend annual discussions with patients once their FEV1 is <50% predicted to allow patients time to become informed about lung transplant. How to integrate caregivers into this discussion is unclear.

Rather than occurring once at the point of care, deliberation is an iterative process in which patients explore what matters most to them when considering medical treatments, often requiring patient collaboration over time with health professionals and their wider social networks. Individuals with CF with all levels of FEV1 report an interest in understanding lung transplant as a potential treatment option. In addition to knowledge gaps about lung transplant identified in a survey of people with CF, investigators found a preparedness gap between how prepared patients feel for the lung transplant decision and how prepared they want to feel. Additionally, the most common patient-endorsed barrier to lung transplant discussions was a worry about being a burden on family and friends after lung transplant. For lung transplant recipients with complex post-operative courses, low social support is associated with increased mortality. Adequate social support is a requirement at all lung transplant programs in the US. Providing support for chronically ill individuals can lead to caregiver burden and burnout. Understanding how to support caregivers of individuals on the lung transplant journey is an important aspect of providing holistic care to people with CF. The CFF recommends routinely measuring caregiver burden using the Brief Assessment Scale for Caregivers (BASC).

Based on prior research, investigators developed a novel lung transplant educational resource that addresses patient-identified knowledge gaps and provides personalized educational content to help people with CF prepare for lung transplant discussions and decisions. The web-based educational resource couples real-life CF patient and caregiver experiences of lung transplant in the form of personal narratives with up-to-date, CF-specific, and guideline-based medical information about lung transplant.

The parent Lung Transplant READY CF 2 study will test the efficacy of the investigator-designed website in a randomized controlled trial (RCT) incorporating mixed methods to assess preparedness for lung transplant discussions among people with CF with FEV1 <50% of predicted, and will explore patient and physician perspectives on the use of the new website for lung transplant education in the era of highly effective CF therapeutics. The overall research objectives for the CARING CF Ancillary RCT will focus on addressing caregivers' education needs, caregiver burden, and understanding the patient-caregiver relationship in decision-making. The central hypothesis is that the investigator-designed website will increase caregivers' preparedness to engage in lung transplant discussions, will lead to greater understanding of the role of caregivers during the transplant journey, and will reduce caregiver burden.

The CARING CF study will be an ancillary RCT. Caregiver participants will take baseline surveys within 3 months of their loved one's enrollment in the parent Lung Transplant READY CF 2 RCT. When the patient participant completes the 3-month study visit in the parent RCT, caregiver participants will repeat surveys and then be randomly assigned 1:1 (stratified by patient's original study arm assignment in parent RCT and patient's baseline report of low social support) to access the investigator-designed website or have no website access for the next three months. Surveys will evaluate knowledge about lung transplant, a Likert scale rating of preparedness for lung transplant discussions, mental health, and caregiver burden (using the BASC). At 3 months after being randomly assigned, there will be a study visit that includes repeated surveys. After completion of the final surveys, all caregiver participants will gain access to the investigator-designed website via individual login to the secure research website. Throughout the 3 months of the randomized portion of the study and for a long-term follow up period of up to 4 years, web analytics will be captured at the individual level to determine caregivers' usage patterns for the research website. Caregivers may be invited to participate in an interview after completion of their final surveys. As part of this ancillary RCT, patient participants who choose to enroll will complete surveys related to their perceived social support at baseline, 3 months and 6 months after their enrollment in the parent RCT and may be invited to participate in an interview with their caregiver.

ELIGIBILITY:
Inclusion Criteria:

* Identified as a caregiver or loved one of an individual with CF enrolled in the Lung Transplant READY CF 2 parent RCT, or
* An individual with CF enrolled in the Lung Transplant READY CF 2 parent RCT

Exclusion Criteria:

* People who are unable to provide informed consent
* Unable to read or understand English or Spanish to complete surveys or access the website (currently only available in English and Spanish)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Brief Assessment Scale for Caregivers (BASC) | Measured at the 3-month and 6-month study visits
  The co-primary endpoint is an intention-to-treat assessment of the difference in caregivers' mean change in Brief Assessment Scale for Caregivers (BASC) in the intervention versus control arms of the study from the 3-month to the 6-month study visit using linear mixed models. The BASC is a validated 14-item measure of caregiver burden and includes subscales that reflect positive personal impact (PPI) and negative personal impact (NPI) of caregiving responsibilities. The BASC includes a 4-point Likert scale (scored 0 to 3), with higher scores indicating more burden, and the overall BASC score is an average of the 14 item scores. The BASC has high internal consistency in caregivers for adults with CF (Cronbach's alpha 0.88 for overall BASC and 0.82 for PPI).
Social Support Effectiveness Questionnaire (SSE-Q) | Measured at the 3-month and 6-month study visits
  A co-primary endpoint is an intention-to-treat assessment of change in patient's Social Support Effectiveness Questionnaire (SSE-Q) from 3 months to 6 months and investigators will compare mean change between patients whose caregivers were randomized to the intervention versus control using linear mixed models. The SSE-Q is a validated 26-item measure of social support with higher scores indicating more effective support. The overall scale ranges from 0 to 80 and each subscale can range from 0 to 20. There are 4 subscales: task support, informational support, emotional support and negative effects of support. The first 15 questions are rated on a 5-point Likert scale and the last questions have yes/no responses. The SSE-Q has not previously been utilized in the CF population.

SECONDARY OUTCOMES:
Confidence-weighted true false knowledge about lung transplant (14-question investigator-designed survey) | Measured at the 3-month and 6-month study visits
  Difference in mean change in confidence-weighted true false (CTF) knowledge score will be measured in the intervention versus control arms of the study using linear mixed models. CTF scoring adds points for certainty in correct responses and deducts points for certainty in incorrect responses. Participants receive +2 points when "sure" about a correct response, +1 if unsure about a correct response, -1 if unsure about an incorrect response and -2 if sure about an incorrect response. For a 14-item knowledge test, the maximum score is +28 and the minimum score is -28, with higher scores indicating more knowledge about lung transplant.
Likert-scale rating of preparedness to discuss lung transplant with their loved one (0-4) | Measured at the 3-month and 6-month study visits
  Likert rating of preparedness to discuss lung transplant with their loved one will be measured at each study visit (0=Don't know, 1= Not at all prepared, 2 = A little prepared, 3 = Moderately prepared, 4 = Very prepared). The intention-to-treat analysis will compare mean change in Likert-scale rating between the intervention and control arms of the study using linear mixed models.
Patient Health Questionnaire (PHQ-8) | Measured at the 3-month and 6-month study visits
  PHQ-8 is a scale that measures symptoms of depression in the prior 2 weeks on a 0-24 scale, with higher scores indicating worsening depression and a score of 10 or higher consistent with a diagnosis of depression. The intention-to-treat analysis will compare mean change in PHQ-8 between the intervention and control arms of the study using linear mixed models. Investigators will also determine the proportion with new PHQ-8 score greater than or equal to 10 in each study arm.
Generalized Anxiety Disorder 7-item (GAD-7) Scale | Measured at the 3-month and 6-month study visits
  GAD-7 is a scale that measures symptoms of anxiety in the prior 2 weeks on a 0-21 scale, with higher scores indicating worsening anxiety and a score of 10 or higher consistent with a diagnosis of generalized anxiety disorder. The intention-to-treat analysis will compare mean change in GAD-7 between the intervention and control arms of the study using linear mixed models. Investigators will also determine the proportion with new GAD-7 score greater than or equal to 10 in each study arm.

OTHER OUTCOMES:
Brief Assessment Scale for Caregivers (BASC): by patient's initial randomization status (intervention or attention control in parent RCT). | Measured at the baseline, 3-month, and 6-month study visits
  Investigators will compare Brief Assessment Scale for Caregivers (BASC) for caregivers of patients initially randomized to intervention in the parent RCT (patient had a chance to learn about lung transplant before their caregiver gained access) versus those randomized to the intervention at the same time as their caregiver (attention control arm initially + caregiver in intervention) versus those whose caregivers had no access to the intervention (patient in either study arm in parent RCT initially + caregiver with no access). All patient participants in the parent RCT will have access to the intervention during the 3-months when the caregivers are randomized to intervention or control. Investigators will assess changes from baseline to 3 months (no caregivers have access to the intervention) and change from 3 to 6 months (caregivers randomized to intervention or control/no access).
Social Support Effectiveness Questionnaire (SSE-Q): by patient's initial randomization status (intervention or attention control in parent RCT). | Measured at the baseline, 3-month, and 6-month study visits
  Investigators will compare Social Support Effectiveness Questionnaire (SSE-Q) for patients initially randomized to intervention in the parent RCT (patient had a chance to learn about lung transplant before their caregiver gained access) versus those randomized to the intervention at the same time as their caregiver (attention control arm initially + caregiver in intervention) versus those whose caregivers had no access to the intervention (patient in either study arm in parent RCT initially + caregiver with no access). All patient participants in the parent RCT will have access to the intervention during the 3-months when the caregivers are randomized to intervention or control. Investigators will assess changes from baseline to 3 months (no caregivers have access to the intervention) and change from 3 to 6 months (caregivers randomized to intervention or control/no access). Higher scores on the SSE-Q indicate more effective support, with a range from 0 to 80.
Assessment of Brief Assessment Scale for Caregivers (BASC): among caregivers of members of communities of concern (low socioeconomic status, Hispanic ethnicity, or Black/Asian/Other race). | Measured at the 3-month and 6-month study visits
  Investigators will assess Brief Assessment Scale for Caregivers (BASC) within the caregivers of patient participants who are members of communities of concern. In an intention-to-treat assessment, investigators will assess the difference in caregivers' mean change in BASC in the intervention versus control arms of the study from the 3-month to the 6-month study visit using linear mixed models, limited to the population of caregivers to patient participants from communities of concern.
Assessment of Social Support Effectiveness Questionnaire (SSE-Q): among members of communities of concern (low socioeconomic status, Hispanic ethnicity, or Black/Asian/Other race). | Measured at the 3-month and 6-month study visits
  Investigators will assess Social Support Effectiveness Questionnaire (SSE-Q) within the cohort of patient participants who are members of communities of concern. In an intention-to-treat assessment, investigators will compare mean change in patient's SSE-Q from 3 months to 6 months between patients whose caregivers were randomized to the intervention versus control using linear mixed models among patient participants who are members of communities of concern. The SSE-Q is a validated 26-item measure of social support with higher scores indicating more effective support. The overall scale ranges from 0 to 80 and each subscale can range from 0 to 20. There are 4 subscales: task support, informational support, emotional support and negative effects of support. The first 15 questions are rated on a 5-point Likert scale and the last questions have yes/no responses. The SSE-Q has not previously been utilized in the CF population.
Assessment of Brief Assessment Scale for Caregivers (BASC): by caregiver gender | Measured at the 3-month and 6-month study visits
  Investigators will assess Brief Assessment Scale for Caregivers (BASC) by caregiver gender, as data in other diseases suggest that women may experience higher levels of caregiver burden and may have a different response to the intervention. In an intention-to-treat assessment, investigators will evaluate the difference in caregivers' mean change in BASC in the intervention versus control arms of the study from the 3-month to the 6-month study visit using linear mixed models, stratified by caregiver gender. The BASC is a validated 14-item measure of caregiver burden and includes subscales that reflect positive personal impact (PPI) and negative personal impact (NPI) of caregiving responsibilities. The BASC includes a 4-point Likert scale (scored 0 to 3), with higher scores indicating more burden, and the overall BASC score is an average of the 14 item scores.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Ramos, MD, MS, Principal Investigator — University of Washington
Locations (1):
- University of Washington Medical Center - Montlake, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) may be shared with other researchers for secondary analyses with the approval of the appropriate Human Subjects Division(s) and the study's principal investigator (PI).
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available after publication of the results of the primary analyses of the study. The data will be available for up to 3 years after the end of the study.
Access Criteria: Qualified researchers with appropriate clinical research training and/or mentorship will be allowed to have access to IPD after approval is obtained from Human Subjects Division(s) and the study PI.

REFERENCES:
- [Background] Ramos KJ, Smith PJ, McKone EF, Pilewski JM, Lucy A, Hempstead SE, Tallarico E, Faro A, Rosenbluth DB, Gray AL, Dunitz JM; CF Lung Transplant Referral Guidelines Committee. Lung transplant referral for individuals with cystic fibrosis: Cystic Fibrosis Foundation consensus guidelines. J Cyst Fibros. 2019 May;18(3):321-333. doi: 10.1016/j.jcf.2019.03.002. Epub 2019 Mar 27. PMID 30926322
- [Background] Hartzler AL, Bartlett LE, Hobler MR, Reid N, Pryor JB, Kapnadak SG, Berry DL, Lober WB, Goss CH, Ramos KJ; Take on Transplant Study Group. Take on transplant: human-centered design of a patient education tool to facilitate informed discussions about lung transplant among people with cystic fibrosis. J Am Med Inform Assoc. 2022 Dec 13;30(1):26-37. doi: 10.1093/jamia/ocac176. PMID 36173364